CLINICAL TRIAL: NCT02945839
Title: Improving Health Outcomes of Migraine Patients Who Present to the Emergency Department
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Significant changes have been made to the protocol.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-00548
Record Dates: First submitted 2016-10-17; First posted 2016-10-26 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Migraine
Keywords: Migraine; emergency department
MeSH Terms: conditions — Migraine Disorders; Emergencies | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acute Treatment+ED-initiated preventive medication +PMR (Active Comparator): All subjects will be discharged on acute migraine therapy (naproxen, triptan) unless there is a contraindication and will also be started on topiramate (25mg/night) with a plan to increase the dose every week by 25 mg up to 100 mg/night. Subjects will receive medicine along with progressive muscle relaxation therapy
  Interventions: Drug: Preventative Medication (PM); Behavioral: Enhanced Usual Care; Behavioral: PMR (progressive muscle relaxation therapy)
- Enhanced Usual Care (EUC) (Active Comparator): Subjects will be given a general education session consisting of basic migraine information such as evidence-based ways to treat migraines: treat early, limit acute medications < 2-3 days/week, and call the primary care physician (PCP) if abortive medications are used more frequently. Any migraine treatment decisions on discharge will be left up to the ED attending. The RC will load the APP onto the subjects' smart phones but the PMR component will be blocked on the version of the APP that they receive. All subjects will be asked to track headache frequency, intensity, and acute medication use on the APP.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Drug: Preventative Medication (PM) — Subjects in the PM group will be given acute migraine medication, preventive medication (topiramate), and the APP with the PMR component. The smartphone app and/or the electronic pill bottles will be used to monitor adherence.
  Other Names: Topiramate
  Arms: Acute Treatment+ED-initiated preventive medication +PMR
Behavioral: Enhanced Usual Care — General Education Class consisting of basic migraine information of basic migraine information such as evidence-based ways to treat migraines: treat early, limit acute medications < 2-3 days/week, and call the primary care physician (PCP) if abortive medications are used more frequently.
Behavioral: PMR (progressive muscle relaxation therapy) — Technique for learning to monitor and control the state of muscular tension
  Arms: Acute Treatment+ED-initiated preventive medication +PMR

SUMMARY:
Collectively, evidence shows that a combination of medication and behavioral therapy is most effective for migraine care. The ED is a critical point of contact with the health care system for many migraine patients; in current practice, it is a missed opportunity to initiate and establish a comprehensive migraine management paradigm. Behavioral headache treatments (e.g., progressive muscle relaxation (PMR), biofeedback, cognitive-behavioral therapy (CBT)) are effective migraine treatment options that are essentially free of side effects. PMR has also been successful as a technique that patients can do independently. Studies have shown that combination pharmacological-behavioral therapy is most effective for migraine treatment.

Several aspects of this study are innovative, including: 1. Initiation of preventive medication in a timely manner for migraineurs who present to the ED. 2. Introduction of PM+PMR in the ED at a time that can serve as a teachable moment. 3. Introduction of a smartphone application-based product (a minimal contact based behavioral therapy) in the ED setting to reduce headache disability, frequency, and intensity.

DETAILED DESCRIPTION:
Investigators will conduct a randomized trial to evaluate the impact of a comprehensive migraine treatment program on the quality of life for migraineurs with frequent and disabling headaches who present to the ED. The intervention (PM+PMR) will combine acute treatment, migraine preventive medication-topiramate, and the APP with PMR. Data from patients in the intervention group will be compared with data from an enhanced usual care (EUC) group to examine the efficacy of the combined treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Meets migraine criteria based on Information in Study Manual or based on Headache expert opinion -4+ migraines a month
* Migraine Disability Assessment (MIDAS) score >5.

Exclusion Criteria:

* Patients who have had Cognitive Behavioral Therapy, Biofeedback or other Relaxation Therapy in the past year;
* Cognitive deficit or other physical problem with the potential to interfere with behavioral therapy; Alcohol or other substance abuse as determined by self-report or prior documentation in the medical record;
* Opioid or barbiturate use 10+ days a month;
* PHQ9 score of severe depression;
* Unable or unwilling to follow a treatment program that relies on written and audio recorded materials;
* Not having a smartphone.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Migraine Disability Assessment Scale (MIDAS) at 3 Months and Baseline | 12 Weeks
  A decrease of 3 points in the MIDAS score corresponds to a one day reduction in headache related disability per month, a clinically meaningful difference.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | 12 Weeks
  PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. A short 4 item scale can be made from questions 2, 4, 5 and 10 of the PSS 10 item scale.
Number of days/week treated with acute medications | 12 Weeks
Number of drug administrations/week for acute medications | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mia Minen, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States